CLINICAL TRIAL: NCT02507115
Title: Text Messaging as a Novel Alcohol Intervention for Community College Students
Acronym: TMAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: Live Inspired, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R21AA021014-01A1 (NIH)
Record Dates: First submitted 2015-07-22; First posted 2015-07-23 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2015-07

CONDITIONS: Alcohol Use
MeSH Terms: conditions — Alcohol Drinking | interventions — 4,4',5'-trimethylazapsoralen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TMAP (Experimental): Alcohol-related Text messages 4 days/week for 6 weeks
  Interventions: Behavioral: TMAP
- Control (Sham Comparator): Motivational Text messages 4 days/week for 6 weeks
  Interventions: Behavioral: Mojo Texts

INTERVENTIONS:
Behavioral: TMAP — Text messages for Alcohol Risk Reduction
  Arms: TMAP
Behavioral: Mojo Texts — Motivational texts not alcohol related
  Arms: Control

SUMMARY:
This project will develop an intervention delivered through text messaging to reduce alcohol consumption and high risk drinking among adults who are enrolled as students in community colleges.

DETAILED DESCRIPTION:
Heavy alcohol use among community college students is a serious problem, leaving students vulnerable to social and health impairment, physical or sexual assault, unintentional injuries, and death. However, there have been limited efforts to research and treat community college students, despite these students comprising nearly 40% of all college students nationwide. Community college students are diverse in ethnicity, age, socioeconomic status, living situation, and employment status. Thus, successful interventions must be sufficiently flexible to apply across a diverse array of individual characteristics and needs. Unfortunately, there is evidence of great unmet need among this group; community college students drive under the influence of alcohol more frequently than students at four-year colleges, and due to lesser time spent on campus, are less available for in-person interventions coordinated at their college. The long-term objective of this research program is to address a gap in the treatment of heavy alcohol use by the community college population. As a first step toward achieving that goal, this R21 application will develop an intervention that is tailored to the needs of community college students and which uses mobile communications platforms that are already used by the vast majority of this population. Taking this approach, the intervention will be mobile, accessible wherever the user is located, and able to be tailored to individual characteristics. The investigators will begin by presenting out initial intervention design to focus groups (4 groups heavy drinking community college students) and obtaining feedback from key informants (advisory board). The investigators will use feedback from these groups to finalize the design and develop a working prototype, and will then pilot the intervention among heavy drinking community college students (N=10) for six weeks to test the usability and acceptability of the prototype intervention. Participants will be interviewed at the end of the program to provide feedback and evaluate their experience with the system, and content experts will again evaluate the prototype using semi-structured interviews. Finally, the investigators will pilot the modified intervention with heaving drinking community college students (N=40) for six weeks. These participants will be randomly assigned to either the intervention program or a standard intervention (print self-help) with a contact-control. Assessments will be conducted at end-of-treatment, and at 3 and 6 months follow up. These data will be used to guide the planning of a full-scale clinical trial to test the efficacy and cost-effectiveness of the intervention in reducing hazardous drinking among community college students

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 28 Community College student Consume at least 4 drinks in one sitting in the past week

Exclusion Criteria:

* none

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number of heavy drinking episodes at six weeks | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The Miriam Hospital- CORO building, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bock BC, Rosen RK, Barnett NP, Thind H, Walaska K, Foster R, Deutsch C, Traficante R. Translating Behavioral Interventions Onto mHealth Platforms: Developing Text Message Interventions for Smoking and Alcohol. JMIR Mhealth Uhealth. 2015 Feb 24;3(1):e22. doi: 10.2196/mhealth.3779. PMID 25714907
- [Result] Bock BC, Barnett NP, Thind H, Rosen R, Walaska K, Traficante R, Foster R, Deutsch C, Fava JL, Scott-Sheldon LA. A text message intervention for alcohol risk reduction among community college students: TMAP. Addict Behav. 2016 Dec;63:107-13. doi: 10.1016/j.addbeh.2016.07.012. Epub 2016 Jul 18. PMID 27450909